CLINICAL TRIAL: NCT04052672
Title: Diet and Exercise Frailty Intervention in Cardiac Device Patients Trial Pilot
Brief Title: Diet and Exercise Frailty Intervention in Cardiac Device Patients
Acronym: DEFINIT-P
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to COVID-19 Pandemic Recruitment was not started
Sponsor: Population Health Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DEFINIT_001
Record Dates: First submitted 2019-07-22; First posted 2019-08-12 (Actual); Last update posted 2022-08-23 (Actual); Status verified 2022-08

CONDITIONS: Frailty; Cardiovascular Diseases
Keywords: Exercise; Nutritional Supplement; Physical Function; Quality of Life; Cardiac Device; Physical Activity; Defibrillators; Pacemakers; Biomarkers
MeSH Terms: conditions — Frailty; Cardiovascular Diseases; Motor Activity | interventions — Exercise; Dietary Supplements

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Randomized Intervention (Active Comparator): The intervention will consist of an exercise intervention, a combination of supervised exercise classes and in home exercises and open label nutritional supplement.
  Interventions: Other: Exercise and Nutritional Supplement
- Randomized - Control (No Intervention): The control will consist of a single group educational session which will include the discussion of general advice on health, exercise and nutrition as well as open label nutritional supplement

INTERVENTIONS:
Other: Exercise and Nutritional Supplement — The intervention consists of exercise (a combination of supervised and in home) as well as a nutritional supplement (a combination of whey protein and creatine).
  Arms: Randomized Intervention

SUMMARY:
DEFINIT-P is a prospective pilot study of frailty in cardiac device recipients, comprised of a registry and randomized control trial. The RCT is a supervised exercise program and nutritional supplement intervention for pre-frail and frail cardiac device participants. The registry will be used to describe all cardiac device recipients, regardless of frailty status.

DETAILED DESCRIPTION:
DEFINIT-P is a single center randomized controlled trial and registry.

This pilot study will determine the feasibility of a larger, multi-center randomized clinical trial which aims to evaluate the efficacy of a supervised exercise program and nutritional supplement program in reversing or preventing progression of frailty in cardiac device recipients.

The future trial would also examine the physiologic effects of exercise and nutritional supplementation to understand their effects on blood biomarker profiles, which will provide insight into potentially targetable mechanisms underlying frailty.

ELIGIBILITY:
Inclusion Criteria

1. Permanent pacemaker recipients OR
2. Implantable cardioverter defibrillator recipients

Exclusion criteria

1. Age <55 years, or
2. Unwilling to consent

Patients will be eligible for the registry but not eligible for the randomized control trial if they fulfill any of:

1. Are non-frail
2. Already undertaking >1 hour per week of dedicated exercise
3. Existing or prior referral for cardiac rehabilitation
4. Moderate or severe heart failure (New York Heart Association class III or IV)
5. Unstable angina
6. Any other medical condition that will prevent exercise participation
7. Dementia, as identified by a Mini-Mental State Examination score <25

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-12-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Rate of identification of eligible patients | 1 year
  The primary outcome will be the number of patients that meet eligibility criteria.
The proportion of eligible patients consenting to participate and randomized | 1 year
  The number of eligible patients that agree to participate in the randomized control trial and the number of eligible patients that consent to participate in the observational trial
The change in the rate of adherence to the trial interventions from baseline to 12 months | 3 months, 6 months, 1 year
  The intervention adherence of both the exercise intervention and nutritional supplement
Barriers and facilitators of adherence to the intervention | 1 year
  The identification of barriers to exercise and nutritional supplement adherence

SECONDARY OUTCOMES:
Frailty biomarker levels | 1 year
  The change in frailty biomarkers (not yet determined) from baseline to 12 months
Physical activity levels as measured by the cardiac device (Permanent pacemaker or Implantable cardioverter defibrillator) | 1 year
  The change in the volume of physical activity as detected by device (hours per day)
Myocardial infarction, stroke, heart failure hospitalization, atrial fibrillation or ventricular tachyarrhythmia | 1 year
  The rate of occurrence of myocardial infarction, stroke, heart failure hospitalization, atrial fibrillation or ventricular tachyarrhythmia
Cardiac device complications | 1 year
  The rate of occurrence of inappropriate defibrillator shocks or lead dislodgement
Injury from a fall or fractures | 1 year
  The rate of occurrence of injury from a fall or fracture

CONTACTS AND LOCATIONS:
Overall Officials: Darryl Leong, PhD. MBBSm, Principal Investigator — McMaster University
Locations (1):
- Hamilton General Hospital, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No